CLINICAL TRIAL: NCT04117607
Title: A Phase 1, Three-Part, Randomized, Double-Blind, Single and Multiple Subcutaneous Dose Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of Rezafungin in Healthy Adult Subjects
Brief Title: Safety and Pharmacokinetics of Rezafungin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped due to the formation of injection site skin nodules.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0088; HHSN272201500007I
Record Dates: First submitted 2019-09-12; First posted 2019-10-07 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2020-06-18

CONDITIONS: Fungal Infection
Keywords: Dose Escalation Study; Double-Blind; Healthy Adult Subjects; Phase 1; Rezafungin; Safety and Pharmacokinetic
MeSH Terms: conditions — Mycoses | interventions — Rezafungin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- BA1 (Experimental): 100 mg (1 injection of 1.0 ml) or maximum tolerated dose (MTD) determined in SAD of Rezafungin administered subcutaneously into the abdomen on Day 1, and 100 mg (250 ml) or MTD of Rezafungin administered via intravenous infusion on Day 22 in an open label manner. n=5.
  Interventions: Drug: Rezafungin
- BA2 (Experimental): 100 mg (250 ml) or maximum tolerated dose (MTD) determined in SAD of Rezafungin administered via intravenous infusion on Day 1, and 100 mg (1 injection of 1.0 ml) or MTD of Rezafungin administered subcutaneously into the abdomen on Day 22 in an open label manner. n=5.
  Interventions: Drug: Rezafungin
- MAD1 (Experimental): 30 mg (1 injection of 0.3 ml) of Rezafungin administered subcutaneously into the abdomen as three doses, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Days 1, 8, and 15 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- MAD2 (Experimental): 60 mg (1 injection of 0.6 ml) of Rezafungin administered subcutaneously into the abdomen as three doses, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Days 1, 8, and 15 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- MAD3 (Experimental): 100 mg (1 injection of 1.0 ml) of Rezafungin administered subcutaneously into alternating abdominal quadrants as three doses, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Days 1, 8, and 15 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- MAD4 (Experimental): 200 mg (2 injections of 1.0 ml) of Rezafungin administered subcutaneously into alternating abdominal quadrants as three doses, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Days 1, 8, and 15 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD1 (Experimental): 1 mg (1 injection of 0.1 ml diluted 1:10 in 5% Dextrose Injection, USP) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=3 (no sentinel dosing), or matching placebo, n=1 (no sentinel dosing), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD2 (Experimental): 10 mg (1 injection of 0.1 ml) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD3 (Experimental): 30 mg (1 injection of 0.3 ml) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD4 (Experimental): 60 mg (1 injection of 0.6 ml) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD5 (Experimental): 100 mg (1 injection of 1.0 ml) of Rezafungin administered subcutaneously into alternating abdominal quadrants as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin
- SAD6 (Experimental): 200 mg (2 injections of 1.0 ml) of Rezafungin administered subcutaneously into alternating abdominal quadrants as a single dose, n=6 (1 sentinel, 5 non-sentinel), or matching placebo, n=2 (1 sentinel, 1 non-sentinel), on Day 1 in a double-blind manner.
  Interventions: Other: Placebo; Drug: Rezafungin

INTERVENTIONS:
Other: Placebo — 5% Dextrose Injection, USP, a sterile, nonpyrogenic solution of dextrose in water for injection. The solution has the osmolarity of 252 mOsmol/L, which is slightly hypotonic. This solution contains no bacteriostat, antimicrobial agent or added buffer.
  Arms: MAD1; MAD2; MAD3; MAD4; SAD1; SAD2; SAD3; SAD4; SAD5; SAD6
Drug: Rezafungin — Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
Drug: Rezafungin — Rezafungin, 200 mg/vial, is a sterile product supplied as a white to pale yellow lyophilized powder in single-dose glass vials for reconstitution with Sterile Water for Injection, United States Pharmacopeia (USP). The reconstituted product is diluted in 0.9% Sodium Chloride Injection, USP for IV infusion. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredients include excipients of mannitol, polysorbate 80, and histidine.
  Arms: BA1; BA2

SUMMARY:
This is a Phase 1, double-blind, placebo-controlled trial in three parts. A single ascending dose (SAD) study in six cohorts receiving a single subcutaneous (SC) dose of 1, 10, 30, 60, 100, or 200 mg of rezafungin; a multiple ascending dose (MAD) study in four cohorts receiving 30 mg x 3 doses, 60 mg x 3 doses, 100 mg x 3 doses, or 200 mg x 3 doses of rezafungin SC with dosing frequency of once every 7 days; and a two-period cross-over bioavailability (BA) study receiving 100 mg of rezafungin. The two period cross-over BA study will be assessed unblinded in two sequences (10 subjects, 100 mg or maximum tolerated dose (MTD) of rezafungin in Part 1); 5 subjects will receive an SC injection of rezafungin in Period 1 followed by an intravenous (IV) infusion of rezafungin in Period 2, and 5 subjects will receive an IV infusion of rezafungin in Period 1 followed by an SC injection of rezafungin in Period 2. Each SAD (except cohort 1) and MAD cohort will contain 8 subjects (6 subjects will receive a SC injection of rezafungin and 2 subjects will receive placebo). Each SAD (except cohort 1) and MAD cohort will be conducted with sentinel dosing. SAD cohort 1 will be comprised of 4 subjects (3:1 rezafungin to placebo) with no sentinel dosing. Parts 2 and 3 of the study will only be conducted after FDA review for safety data and PK data from all subjects participating in Part 1; Part 3 may be run in parallel with the first cohort (Cohort 7) of Part 2. Individuals in the SAD cohorts will participate for approximately 58 days, including up to 28 days for screening and 30 days for dosing and follow-up (FU). Individuals in the MAD cohorts will participate for approximately 73 days, including up to 28 days for screening and 45 days for dosing and FU. Individuals in the BA cohorts will participate for approximately 80 days, including up to 28 days for screening and 52 days for dosing and FU. The study will have a duration of approximately 30 months. The primary objectives are to determine the: 1) safety and tolerability of single ascending SC doses (SAD) of rezafungin; 2) safety and tolerability of multiple ascending SC doses (MAD) of rezafungin; and 3) pharmacokinetic (PK) profile in plasma of rezafungin in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled trial in three parts. A single ascending dose (SAD) study in six cohorts receiving a single subcutaneous (SC) dose of 1, 10, 30, 60, 100, or 200 mg of rezafungin; a multiple ascending dose (MAD) study in four cohorts receiving 30 mg x 3 doses, 60 mg x 3 doses, 100 mg x 3 doses, or 200 mg x 3 doses of rezafungin SC with dosing frequency of once every 7 days; and a two-period cross-over bioavailability (BA) study receiving 100 mg of rezafungin. The two period cross-over BA study will be assessed unblinded in two sequences (10 subjects, 100 mg or maximum tolerated dose (MTD) of rezafungin in Part 1); 5 subjects will receive an SC injection of rezafungin in Period 1 followed by an intravenous (IV) infusion of rezafungin in Period 2, and 5 subjects will receive an IV infusion of rezafungin in Period 1 followed by an SC injection of rezafungin in Period 2. Each SAD (except cohort 1) and MAD cohort will contain 8 subjects (6 subjects will receive a SC injection of rezafungin and 2 subjects will receive placebo). Each SAD (except cohort 1) and MAD cohort will be conducted with sentinel dosing. SAD cohort 1 will be comprised of 4 subjects (3:1 rezafungin to placebo) with no sentinel dosing. Parts 2 and 3 of the study will only be conducted after FDA review for safety data and PK data from all subjects participating in Part 1; Part 3 may be run in parallel with the first cohort (Cohort 7) of Part 2. Individuals in the SAD cohorts will participate for approximately 58 days, including up to 28 days for screening and 30 days for dosing and follow-up (FU). Individuals in the MAD cohorts will participate for approximately 73 days, including up to 28 days for screening and 45 days for dosing and FU. Individuals in the BA cohorts will participate for approximately 80 days, including up to 28 days for screening and 52 days for dosing and FU. The study will have a duration of approximately 30 months. The primary objectives are to determine the: 1) safety and tolerability of single ascending SC doses (SAD) of rezafungin; 2) safety and tolerability of multiple ascending SC doses (MAD) of rezafungin; and 3) pharmacokinetic (PK) profile in plasma of rezafungin in healthy adult subjects. The secondary objective is to evaluate the BA of rezafungin when administered by SC injection relative to IV infusion in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 45 years, inclusive.
2. Willing and able to provide written informed consent and authorization for use of protected health information.
3. Willing and able to comply with protocol requirements, instructions, and protocol-stated restrictions (including confinement to the Clinical Research Unit) and is likely to complete the study as planned.
4. Males must be vasectomized or agree to use barrier contraception (condom with spermicide) from first dose of study drug until at least 18 weeks following the last dose of study drug.
5. Males must agree to refrain from sperm donation from first dose of investigational product (IP) through at least 18 weeks after last dose of IP.
6. Females are eligible if they are of non-childbearing potential* or if they use a highly effective** method of contraception for 30 days prior to dosing and for a minimum of 30 days after dosing.

   *Non-childbearing potential is defined as: Pre-menopausal with documentation of irreversible surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, or bilateral salpingectomy (but not tubal ligation alone); or, Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with Follicle Stimulating Hormone (FSH) levels > / = 40 mIU/mL at Screening.

   **A highly effective contraceptive method is, defined by < 1 percent failure rate that is not affected by user adherence, include surgical sterilization and long-acting reversible contraception (LARC). LARC comes in three forms: progestin-releasing subdermal implants (Nexplanon and Implanon [Merck]); copper intrauterine devices (IUD) (ParaGard [Teva]); and levonorgestrel-releasing IUDs (Mirena [Bayer], Skyla [Bayer], and Liletta [Allergan/Medicines360]. Subjects must use one of these three methods.
7. Subject is in good health as deemed by the Investigator*,**.

   * Good health is defined by the absence of any medical condition described in the exclusion criteria in a subject who undergoes a medical history, with a normal complete physical examination including resting vital signs, and screening safety laboratory testing.

     * If the subject has an active, ongoing medical condition, the condition cannot meet any of the following criteria: 1) first diagnosed within 3 months of enrollment; 2) is worsening in terms of clinical outcome in last 6 months; or 3) involves need for medication that may pose a risk to subject's safety or significantly impede assessment of adverse events if they participate in the study.
8. Subjects with a body mass index (BMI) (weight in kg divided by height in m, squared) between 18.5 and/or 35.0 kg/m^2, inclusive, and a minimum weight of 50 kg.
9. Subjects must refrain from strenuous physical activity that could cause muscle aches or injury, including contact sports, at any time from screening until completion of the trial.
10. Subjects must refrain from over-the-counter and prescription medications* and nutritional supplements within 14 days before first study drug administration, and until after the final study visit.

    *Except for hormonal contraceptives, acetaminophen, or ibuprofen.
11. Subject has adequate venous access for blood collection.

Exclusion Criteria:

1. History of any hypersensitivity or allergic reaction to echinocandins or excipients (mannitol, polysorbate 80, histidine) of the rezafungin for injection and rezafungin for infusion formulations.
2. Subjects presenting with a clinically significant condition*.

   *Subjects with any of the following must not be included into the study: clinically significant oncologic, infectious, cardiovascular, pulmonary, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, immunologic, renal, psychiatric, or other condition that in the opinion of the Investigator would preclude the safe participation of the subject in the study or would prevent the subject from meeting the study requirements.
3. Any condition that in the opinion of the Investigator could significantly impact drug absorption, distribution, or elimination.
4. Symptoms of acute illness or chronic disease within 14 days of initial dosing.
5. Positive screen for hepatitis B virus surface antigen, hepatitis C virus antibody, or Human Immunodeficiency Virus (HIV) antibody.
6. Subjects with clinical laboratory values outside the site reference ranges* prior to initial dosing.

   *Clinical laboratory values outside the site reference ranges, if considered by the site investigator to be clinically insignificant, are acceptable if not exceeding Grade 1 severity. One repeat of lab testing is allowed to make this determination during screening.
7. Abnormal Electrocardiograms (ECGs).
8. Female subject of childbearing potential who is pregnant*, lactating, or planning to become pregnant during the study period or at least 30 days after the final dose of study product.

   *Having a positive serum pregnancy test at the Screening Visit or any other specified time point prior to the dose of study product.
9. Received any prescription medications (except for hormonal contraceptives) within 14 days before first study drug administration.
10. Received any non-prescription medications, vitamins, herbal or dietary supplements* within 14 days of initial dosing, unless prior approval is granted by both the Investigator and the Sponsor.

    *Excluded from this list is intermittent use of acetaminophen at doses of < / = 2 g/day or ibuprofen < / = 1200 mg/day. However, acetaminophen only is accepted to treat AEs for pain (ie. headaches) during in-clinic stay.
11. Current smoker or tobacco* use within 90 days prior to screening or while a subject is enrolled in the study.

    *Tobacco use includes vaping, smoking tobacco, the use of snuff and chewing tobacco, and other nicotine or nicotine-containing products
12. History of illicit/illegal drug use prior to dosing or while a subject is enrolled in the study* or reports an alcohol or substance abuse problem** within 6 months of dosing.

    *A urine drug test will be performed at screening and upon admission to the Clinical Research Unit (CRU). Drug screen includes amphetamines, barbiturates, cocaine, opiates, cannabinoids, phencyclidine, and benzodiazepines.

    **Inclusive of vaping of non-nicotine products.
13. Consumed foods or beverages containing alcohol or xanthines/caffeine*,**:

    *Alcohol: < / = 48 hours before the first study drug administration, until discharge.

    **Xanthines/caffeine: < / = 24 hours before the first study drug administration, until discharge.
14. Received any live or killed vaccines or immunoglobulins within 14 days of dosing.
15. Donated blood or blood products or experienced significant blood loss within 60 days of dosing.
16. Received a blood transfusion within 14 days of dosing.
17. Previous participation in this trial, any other rezafungin trial, or any trial* within 28 days of dosing. Plans to enroll in another clinical trial**.

    *Includes trials that have a study intervention such as a drug, biologic, or device.

    **Includes trials that could interfere with safety assessment of the investigational product at any time during the study period.
18. The PI considers that the subject should not participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Services Clinical Research Unit, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included healthy male and females aged 18-45 years (inclusive). Participants were recruited from the local community to ensure that male, female, and minorities (African American, Native American, Asian, and Hispanics) were represented in the enrolled population. Participants were enrolled between 04DEC2019 and 11MAR2020.
Groups:
- SAD1: 1 mg (1 injection of 0.1 mL diluted 1:10 in 5% Dextrose Injection, USP) of Rezafungin administered subcutaneously into the abdomen as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD2: 10 mg (1 injection of 0.1 mL) of Rezafungin administered subcutaneously into the abdomen as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD3: 30 mg (1 injection of 0.3 mL) of Rezafungin administered subcutaneously into the abdomen as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD4: 60 mg (1 injection of 0.6 mL) of Rezafungin administered subcutaneously into the abdomen as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD5: 100 mg (1 injection of 1.0 mL) of Rezafungin administered subcutaneously as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD6: 200 mg (2 injections of 1.0 mL) of Rezafungin administered subcutaneously into the same abdominal quadrant (separated by approximately 5 cm) as a single dose, on Day 1 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- SAD Placebo: Placebo participants across all SAD cohorts: 1 mg (1 injection of 0.1 mL diluted 1:10 in 5% Dextrose Injection, USP), 10 mg (1 injection of 0.1 ml), 30 mg (1 injection of 0.3 ml), 60 mg (1 injection of 0.6 ml), 100 mg (1 injection of 1 ml), or 200 mg (2 injections of 1 ml) of matching placebo administered subcutaneously as a single dose in a double-blind manner on Day 1 in a double-blind manner.
  The 200 mg dose injections will be administered in the same abdominal quadrant, separated by approximately 5 cm.
  Placebo: 5% Dextrose Injection, USP, a sterile, nonpyrogenic solution of dextrose in water for injection. The solution has the osmolarity of 252 mOsmol/L, which is slightly hypotonic. This solution contains no bacteriostat, antimicrobial agent or added buffer.
- MAD1: 30 mg (1 injection of 0.3 mL) of Rezafungin administered subcutaneously into the abdomen as three doses, with each dose administered in a different quadrant (3 quadrants total), on Days 1, 8, and 15 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- MAD2: 60 mg (1 injection of 0.6 mL) of Rezafungin administered subcutaneously into the abdomen as three doses, with each dose administered in a different quadrant (3 quadrants total), on Days 1, 8, and 15 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- MAD3: 100 mg (1 injection of 1.0 mL) of Rezafungin administered subcutaneously into the abdomen as as three doses, with each dose administered in a different quadrant (3 quadrants total), on Days 1, 8, and 15 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- MAD4: 200 mg (2 injections of 1.0 mL) of Rezafungin administered subcutaneously into the abdomen as three doses, each injection will be administered in the same quadrant (separated by approximately 5 cm) and each separate dose will be administered into different abdominal quadrants (3 quadrants total), on Days 1, 8, and 15 in a double-blind manner.
  Rezafungin: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
- MAD Placebo: Placebo participants across all MAD cohorts: 30 mg (1 injection of 0.3 mL), 60 mg (1 injection of 0.6 ml), 100 mg (1 injection of 1.0 ml), 200 mg (2 injections of 1.0 ml), of matching placebo administered subcutaneously as three doses on Days 1, 8, and 15 in a double-blind manner. The 200 mg dose injections will be administered in the same abdominal quadrant, separated by approximately 5 cm. Each dose will be administered in a different quadrant (3 quadrants total).
  Placebo: 5% Dextrose Injection, USP, a sterile, nonpyrogenic solution of dextrose in water for injection. The solution has the osmolarity of 252 mOsmol/L, which is slightly hypotonic. This solution contains no bacteriostat, antimicrobial agent or added buffer.
- BA 1: 100 mg (1 injection of 1.0 mL) or maximum tolerated dose (MTD) of Rezafungin, determined in part 1 of the study (SAD), administered subcutaneously into the abdomen on Day 1, and 100 mg (250 mL) or MTD of Rezafungin administered via intravenous infusion over 60 minutes on Day 22 in an open label manner.
  Rezafungin for subcutaneous use: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
  Rezafungin for intravenous infusion: Rezafungin, 200 mg/vial, is a sterile product supplied as a white to pale yellow lyophilized powder in single-dose glass vials for reconstitution with Sterile Water for Injection, United States Pharmacopeia (USP). The reconstituted product is diluted in 0.9% Sodium Chloride Injection, USP for IV infusion. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredients include excipients of mannitol, polysorbate 80, and histidine.
- BA 2: 100 mg (250 mL) or maximum tolerated dose (MTD) of Rezafungin, determined in part 1 of the study (SAD), administered via intravenous infusion over 60 minutes on Day 1, and 100 mg (1 injection of 1.0 mL) or MTD of Rezafungin administered subcutaneously into the abdomen on Day 22 in an open label manner.
  Rezafungin for subcutaneous use: Rezafungin, 100 mg/mL, is a sterile liquid product supplied in single-dose vials containing 1.0 mL of extractable volume. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredient is mannitol.
  Rezafungin for intravenous infusion: Rezafungin, 200 mg/vial, is a sterile product supplied as a white to pale yellow lyophilized powder in single-dose glass vials for reconstitution with Sterile Water for Injection, United States Pharmacopeia (USP). The reconstituted product is diluted in 0.9% Sodium Chloride Injection, USP for IV infusion. The active pharmaceutical ingredient is rezafungin acetate, a water-soluble amorphous acetate salt. The inactive ingredients include excipients of mannitol, polysorbate 80, and histidine.
Period: Overall Study
Arm/Group | SAD1 | SAD2 | SAD3 | SAD4 | SAD5 | SAD6 | SAD Placebo | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo | BA 1 | BA 2
Started | 3 | 7 | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 4 | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.) | 0 (The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.)
Received Study Product | 3 | 6 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed All PK Blood Draws | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 6 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Early Termination | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of subjects randomized.
Groups:
- SAD1: 1 mg (1 injection of 0.1 mL diluted 1:10 in 5% Dextrose Injection, USP) of Rezafungin administered subcutaneously.
- SAD2: 10 mg (1 injection of 0.1 mL) of Rezafungin administered subcutaneously.
- SAD Placebo: Placebo participants across all SAD cohorts given matching placebo administered subcutaneously as a single dose in a double-blind manner.
- Total: Total of all reporting groups
Arm/Group | SAD1 | SAD2 | SAD Placebo | Total
Number analyzed (Participants) | 3 | 7 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (2.1) | 33.6 (6.5) | 33.8 (7.5) | 33.6 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 3 | 6 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 1 | 5 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 1 | 4
  White | 2 | 3 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 174.73 (8.84) | 177.74 (5.77) | 172.1 (6.15) | 175.49 (6.52)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 85.9 (13.75) | 88.13 (17) | 77.23 (18.67) | 84.54 (16.33)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.97 (1.72) | 27.74 (4.18) | 25.85 (4.23) | 27.25 (3.67)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 2
Description: Laboratory parameters and associated thresholds include albumin <=3.4 g/dL, glucose <= 69 mg/dL or >=106 mg/dL, blood urea nitrogen (BUN) >= 21 mg/dL, potassium >=5.2 mEq/L or <=3.4 mEq/L, calcium < 8.7 mg/dL or >=10.3 mg/dL, sodium <=132 mEq/L or >=144 mEq/L, total protein <=5.9 g/dL, creatinine >=1.3 mg/dL (male) or >= 1.0 mg/dL (female), creatine phosphokinase >= 309 U/L, phosphorus <=2.4 mg/dL, alkaline phosphatase >= 131 IU/L (males) or >= 106 IU/L (female), aspartate aminotransferase >= 40 U/L (male) or >= 32 U/L (female), alanine aminotransferase >=41 U/L (male) or >= 33 U/L (female), and total bilirubin >=106 mg/dL. If a clinical chemistry laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 1 | 0
  Alanine Aminotransferase, Increase | 0 | 1 | 0
  Glucose, Increase | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 7
Description: as for outcome 1
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 0 | 2 | 1
  Potassium, Increase | 0 | 1 | 0
  Calcium, Increase | 0 | 0 | 1
  Alanine Aminotransferase, Increase | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 30
Description: as for outcome 1
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 0 | 3 | 0
  Alanine Aminotransferase, Increase | 0 | 3 | 0

4. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results for Multiple Ascending Dose (MAD)
Description: as for outcome 1
Time Frame: Day 2 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Groups:
- MAD1: 30 mg (1 injection of 0.3 mL) of Rezafungin administered subcutaneously.
- MAD2: 60 mg (1 injection of 0.6 mL) of Rezafungin administered subcutaneously.
- MAD3: 100 mg (1 injection of 1.0 mL) of Rezafungin administered subcutaneously.
- MAD4: 200 mg (2 injections of 1.0 mL) of Rezafungin administered subcutaneously.
- MAD Placebo: Placebo participants across all MAD cohorts given matching placebo administered subcutaneously.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 2
Description: Laboratory parameters and associated thresholds for adverse events include hemoglobin <= 12.2 g/dL (male) or <= 10.8 g/dL (female), hematocrit <= 36.1 % (male) or <= 32.6 % (female), red blood cell (RBC) count <= 4.1 x 10^6/uL (male) or <= 3.7 x 10^6/uL (female), white blood cell (WBC) count >= 9,001 cell/mm3 or <= 2,499 cell/mm3 (African American Males) or >= 11,001 cell/mm3 or <= 2,499 cell/mm3 (African American Females) or >= 10,001 cell/mm3 or <= 3,999 cell/mm3 (all others), neutrophil count <= 1,299 cell/mm3 (African Americans) or <= 1,699 cell/mm3 (all others), lymphocyte count <= 799 cell/mm3, monocyte count >= 1001 cell/mm3, eosinophil count >= 871 cell/mm3, basophil count >= 101 cell/mm3, and platelet count <= 149 x 10^3/mm3. If a result met the threshold for an AE at baseline, subsequent results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 1 | 1
  White Blood Cell Count, Decrease | 0 | 0 | 1
  White Blood Cell Count, Increase | 0 | 1 | 0
  Neutrophil Count, Decrease | 1 | 0 | 0
  Monocyte Count, Increase | 0 | 1 | 0
  Basophil Count, Increase | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 7
Description: as for outcome 5
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 0 | 1 | 1
  White Blood Cell Count, Decrease | 0 | 0 | 1
  White Blood Cell Count, Increase | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results for Single Ascending Dose (SAD) on Day 30
Description: as for outcome 5
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 2 | 0 | 0
  Neutrophil Count, Decrease | 1 | 0 | 0
  Eosinophil Count, Increase | 1 | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results for Multiple Ascending Dose (MAD)
Description: as for outcome 5
Time Frame: Day 2 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 2
Description: Laboratory parameters include prothrombin time (PT), activated partial prothrombin time (PTT), and prothrombin international normalized ratio (INR). Thresholds for adverse events were considered as PT >= 11.1 s (before 23DEC2019) or >= 11.6 s (on or after 23DEC2019), PTT >= 34.1 s (before 23DEC2019) or >= 30.1 (on or after 23DEC2019), INR >= 1.2. If a coagulation laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 7
Description: as for outcome 9
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 30
Description: as for outcome 9
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results for Multiple Ascending Dose (MAD)
Description: as for outcome 9
Time Frame: Day 2 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 2
Description: Laboratory parameters include protein, glucose, and occult blood. Thresholds for adverse events were considered as protein >= 1+, glucose >= 1+, and occult blood >= 5 (before 23DEC2019) or >=3 (on or after 23DEC2019). If a urinalysis laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 7
Description: as for outcome 13
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 0 | 1 | 0
  Protein by Dipstick | 0 | 1 | 0

15. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results for Single Ascending Dose (SAD), Day 30
Description: as for outcome 13
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results for Multiple Ascending Dose (MAD)
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Laboratory parameters include protein, glucose, and occult blood. Thresholds for adverse events were considered as protein >= 1+, glucose >= 1+, and occult blood >= 5 (before 23DEC2019) or >=3 (on or after 23DEC2019). If a urinalysis laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 2 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormal ECG Toxicity Results for Single Ascending Dose (SAD), Day 1
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. ECG parameters include PR interval and QTcF interval. Thresholds for adverse events were considered as PR interval >= 0.21 sec, a type II 2nd degree AV block, or ventricular pause >3 sec and QTcF interval >= 450 msec or >= 30 msec above baseline. If an ECG value met the threshold for an AE at baseline, subsequent safety ECG results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Abnormal ECG Toxicity Results for Single Ascending Dose (SAD), Day 7
Description: as for outcome 17
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Abnormal ECG Toxicity Results for Single Ascending Dose (SAD), Day 30
Description: as for outcome 17
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

20. Primary Outcome: Number of Participants With Abnormal ECG Toxicity Results for Multiple Ascending Doses (MAD)
Description: This table includes the maximum severity experienced over all post-baseline time points. ECG parameters include PR interval and QTcF interval. Thresholds for adverse events were considered as PR interval >= 0.21 sec, a type II 2nd degree AV block, or ventricular pause >3 sec and QTcF interval >= 450 msec or >= 30 msec above baseline. If an ECG value met the threshold for an AE at baseline, subsequent safety ECG results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Number of Participants With Abnormal Physical Exams for Single Ascending Dose (SAD), Day 1
Description: Physical examination includes general appearance; head, eyes, nose and throat; neck; chest and lungs; cardiovascular system, abdomen, musculoskeletal system, lymph nodes, extremities/skin, and neurological system.
Time Frame: Day 1
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
participants
  Any Parameter | 0 | 1 | 0
  Extremities/skin | 0 | 1 | 0

22. Primary Outcome: Number of Participants With Abnormal Physical Exams for Single Ascending Dose (SAD), Day 2
Description: as for outcome 21
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
participants
  Any Parameter | 0 | 6 | 0
  Extremities/skin | 0 | 6 | 0

23. Primary Outcome: Number of Participants With Abnormal Physical Exams for Single Ascending Dose (SAD), Day 4
Description: as for outcome 21
Time Frame: Day 4
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
participants
  Any Parameter | 0 | 5 | 0
  Extremities/skin | 0 | 5 | 0

24. Primary Outcome: Number of Participants With Abnormal Physical Exams for Single Ascending Dose (SAD), Day 7
Description: as for outcome 21
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
participants
  Any Parameter | 0 | 1 | 0
  Extremities/skin | 0 | 1 | 0

25. Primary Outcome: Number of Participants With Abnormal Physical Exams for Single Ascending Dose (SAD), Day 30
Description: as for outcome 21
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
participants
  Any Parameter | 0 | 2 | 0
  Extremities/skin | 0 | 2 | 0

26. Primary Outcome: Number of Participants With Abnormal Physical Exams for Multiple Ascending Dose (MAD)
Description: as for outcome 21
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into these groups.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 1, 15 Minutes Post-dose
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Vital sign parameters include systolic blood pressure (BP), diastolic BP, heart rate, respiratory rate, and temperature. Thresholds for abnormal vital signs were considered as systolic BP >= 141 mmHg or <= 89 mmHg, diastolic BP >= 91 mmHg, heart rate <= 54 bpm (baseline >= 60 bpm) or <=50 (baseline < 60 bpm) or >= 101 bpm, respiratory rate >= 23 breaths per minute, and temperature >= 38.0 degrees Celsius. If a vital sign result met the threshold for an AE at baseline, subsequent vital sign results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1, 15 minutes post-dose
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

28. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 1, 1 Hour Post-dose
Description: as for outcome 27
Time Frame: Day 1, 1 hour post-dose
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 0 | 2 | 0
  Heart Rate, Decrease | 0 | 2 | 0

29. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 1, 2 Hours Post-dose
Description: as for outcome 27
Time Frame: Day 1, 2 hours post-dose
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

30. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 2
Description: as for outcome 27
Time Frame: Day 2
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 0 | 0
  Heart Rate, Decrease | 1 | 0 | 0

31. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 4
Description: as for outcome 27
Time Frame: Day 4
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 0 | 0
  Heart Rate, Decrease | 1 | 0 | 0

32. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 7
Description: as for outcome 27
Time Frame: Day 7
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 0 | 0
  Heart Rate, Decrease | 1 | 0 | 0

33. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 14
Description: as for outcome 27
Time Frame: Day 14
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 0 | 0
  Heart Rate, Decrease | 1 | 0 | 0

34. Primary Outcome: Number of Participants With Abnormal Vital Signs for Single Ascending Dose (SAD), Day 30
Description: as for outcome 27
Time Frame: Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Parameter | 1 | 0 | 0
  Heart Rate, Decrease | 1 | 0 | 0

35. Primary Outcome: Number of Participants With Abnormal Vital Signs for Multiple Ascending Dose (MAD)
Description: as for outcome 27
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this group.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

36. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) for Single Ascending Dose (SAD)
Description: Number of participants with an AE are summarized by MedDRA System Organ Class (SOC) and severity. If a condition was present at screening it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 30.
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any SOC | 3 | 6 | 2
  Investigations | 2 | 5 | 2
  Cardiac disorders | 0 | 2 | 0
  General disorders and administration site conditions | 0 | 2 | 0

37. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) for Multiple Ascending Dose (MAD)
Description: Number of participants with an AE are summarized by MedDRA System Organ Class (SOC). Each subject was counted once per SOC. If a condition was present at screening, it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any MAD cohorts.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

38. Primary Outcome: Number of Unsolicited Adverse Events Reported for Single Ascending Dose (SAD)
Description: The total number of unsolicited AE events reported summarized by MedDRA System Organ Class (SOC). If a condition was present at screening it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 30.
Population: Safety population: All participants that received any amount of study product.
Measure: Number; unit: AE events
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
AE events
  Any SOC | 8 | 14 | 2
  Investigations | 4 | 8 | 2
  Cardiac Disorders | 0 | 2 | 0
  General disorders and administration site conditions | 0 | 2 | 0

39. Primary Outcome: Number of Unsolicited Adverse Events Reported for Multiple Ascending Dose (MAD)
Description: as for outcome 38
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any MAD cohorts.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

40. Primary Outcome: Number of Participants With at Least One Severe Adverse Event (SAE) for Single Ascending Dose (SAD)
Description: The number of participants who reported at least one SAE. SAEs include any AE that resulted in death, a life-threatening event, an inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants | 0 | 0 | 0

41. Primary Outcome: Number of Participants With at Least One Severe Adverse Event (SAE) for Multiple Ascending Dose (MAD)
Description: as for outcome 40
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any MAD cohorts.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

42. Primary Outcome: Number of Participants With Solicited Local Reactogenicity Symptom(s) for Single Ascending Dose (SAD)
Description: The number of participants who experienced solicited local reactogenicity events (injection site evaluation), summarized by symptom. Specified solicited events include pain, tenderness, pruritus, ecchymosis, erythema, induration, nodule, ulcer, healed, and scar. Thresholds for measurement grades of solicited local reactogenicity events were considered as ecchymosis >= 25 mm, erythema >=25 mm, induration >=25 mm, nodule >=25 mm, ulcer >=1 mm. For functional grades of solicited local reactogenicity events, the threshold for tenderness was considered as discomfort only to the touch or worse. For ecchymosis, erythema, induration, nodule, or ulcer thresholds for functional grade was interference with daily activity or worse, or any measurement over 1mm.
Time Frame: Day 1 through Day 30
Population: Safety population: All participants that received any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD1 | SAD2 | SAD Placebo
Number analyzed (Participants) | 3 | 6 | 3
Participants
  Any Symptom | 1 | 6 | 0
  Pain | 1 | 2 | 0
  Tenderness | 0 | 4 | 0
  Pruritus | 0 | 1 | 0
  Ecchymosis, Functional Grade | 0 | 2 | 0
  Ecchymosis, Measurement Grade | 0 | 1 | 0
  Induration/Swelling, Functional Grade | 0 | 1 | 0
  Induration/Swelling, Measurement Grade | 0 | 1 | 0
  Erythema, Functional Grade | 0 | 6 | 0
  Erythema, Measurement Grade | 0 | 6 | 0
  Nodule, Functional Grade | 0 | 5 | 0
  Nodule, Measurement Grade | 0 | 4 | 0
  Ulceration, Functional Grade | 0 | 0 | 0
  Ulceration, Measurement Grade | 0 | 0 | 0

43. Primary Outcome: Number of Participants With Solicited Local Reactogenicity Symptom(s) for Multiple Ascending Dose (MAD)
Description: as for outcome 42
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into this cohort.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

44. Primary Outcome: Rezafungin Concentrations in Plasma, SAD 10 mg Dose Group Concentrations of Rezafungin in Plasma Samples
Description: Mean and standard deviation of rezafungin concentrations in plasma from the SAD 10 mg Dose Group by nominal time point (0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, 696 h (post-dose)).
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed one full 10 mg rezafungin dose, as randomized and according to cohort; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD2
Number analyzed (Participants) | 6
ng/mL
  0 h | 0 (0)
  0.5 h | 0 (0)
  1 h | 0 (0)
  2 h | 8.983 (7.386)
  4 h | 21.5 (7.954)
  6 h | 28.68 (9.949)
  8 h | 36.35 (13.62)
  12 h | 45.9 (17.56)
  24 h | 70.87 (23.52)
  48 h | 97.75 (27.35)
  96 h | 101.8 (28.3)
  144 h | 99.9 (30.15)
  312 h | 49.5 (15.06)
  696 h: number analyzed (Participants) | 5
  696 h | 14.52 (3.594)

45. Primary Outcome: Rezafungin PK Parameter (Cmax) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the Cmax (ng/mL) PK parameter estimated from the rezafungin plasma concentration-time data.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD2
Number analyzed (Participants) | 6
ng/mL | 108.3 (29.5)

46. Primary Outcome: Rezafungin PK Parameters (Tmax and t 1/2) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the Tmax (h) and t 1/2 (h) PK parameters were estimated from the rezafungin plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 3.0 half-lives, and includes at least 3 timepoints after tmax.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed 10 mg rezafungin dose as randomized; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
  t 1/2 was inestimable for all subjects due to not meeting the specified lambda z acceptance criteria.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SAD2
Number analyzed (Participants) | 6
h
  Tmax | 120 (40.16)
  t1/2: number analyzed (Participants) | 0

47. Primary Outcome: Rezafungin PK Parameters (AUC 0-last and AUC 0-inf ) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the AUC 0-last (h*ng/mL) and AUC 0-inf (h*ng/mL) PK parameters were estimated from the rezafungin plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 3.0 half-lives, and includes at least 3 timepoints after tmax.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed 10 mg rezafungin dose as randomized; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
  AUC 0-inf was inestimable for all subjects due to not meeting the specified lambda z acceptance criteria.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAD2
Number analyzed (Participants) | 6
h*ng/mL
  AUC 0-last | 33950 (9989)
  AUC 0-inf: number analyzed (Participants) | 0

48. Primary Outcome: Rezafungin PK Parameter (Lambda z) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the lambda z (1/h) PK parameter was estimated from the rezafungin plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 3.0 half-lives, and includes at least 3 timepoints after tmax.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed 10 mg rezafungin dose as randomized; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
  Lambda z was inestimable for all subjects due to not meeting the specified lambda z acceptance criteria.
Arm/Group | SAD2
Number analyzed (Participants) | 0

49. Primary Outcome: Rezafungin PK Parameter (CL/F) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the CL/F (L/h) PK parameter was estimated from the rezafungin plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 3.0 half-lives, and includes at least 3 timepoints after tmax.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed 10 mg rezafungin dose as randomized; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
  CL/F was inestimable for all subjects due to not meeting the specified lambda z acceptance criteria.
Arm/Group | SAD2
Number analyzed (Participants) | 0

50. Primary Outcome: Rezafungin PK Parameter (Vz/F) in Plasma, SAD 10 mg Dose Group
Description: Mean and standard deviation (SD) of the Vz/F (L) PK parameter was estimated from the rezafungin plasma concentration-time data using Phoenix WinNonlin Non-compartmental Analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 3.0 half-lives, and includes at least 3 timepoints after tmax.
Time Frame: 0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h, 48 h, 96 h, 144 h, 312 h, and 696 h post-dose
Population: PK Analysis Subset: All participants who completed 10 mg rezafungin dose as randomized; had at least one post-dose plasma sample with a measurable rezafungin concentration from which at least a subset of the designated PK parameters could be determined; and completed the PK part of the trial without any protocol violations that were likely to affect the PK results.
  Vz/F was inestimable for all subjects due to not meeting the specified lambda z acceptance criteria.
Arm/Group | SAD2
Number analyzed (Participants) | 0

51. Primary Outcome: Rezafungin Concentrations in Plasma Samples, Multiple Ascending Dose (MAD)
Description: Mean and standard deviation of rezafungin concentrations in plasma from the SAD 10 mg Dose Group by nominal time point (0 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, and 12 h on Days 1 and 15, 24 h post-dose on Days 2 and 16, 48 h post-dose on Days 3 and 17; at 1 h and 4 h post-dose on Day 8; at 72 h post-dose on Days 4, 11, and 18; at 96 hours post-dose on Days 5, 12, and 19; at 120 h post-dose on Days 6, 13, and 20; at 144 h post-dose on Days 7, 14, and 21; on Days 30 and 45 post-dose)
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any of the MAD cohorts.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

52. Primary Outcome: Rezafungin PK Parameters in Plasma, Multiple Ascending Dose (MAD)
Description: Mean and standard deviation (SD) of PK parameters estimated from the rezafungin plasma concentration-time data. PK Parameters include Cmax (ng/nL), Tmax (h), AUC 0-last (h*ng/mL), AUC 0-inf (h*ng/mL), lambda z (1/h), t 1/2 (h), CL/F (L/h), Vz/F (L).
Time Frame: Day 1 through Day 45
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any of the MAD cohorts.
Arm/Group | MAD1 | MAD2 | MAD3 | MAD4 | MAD Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Bioavailability (BA) of Rezafungin in BA Cohorts
Description: BA is calculated as the ratio of the area under the curve (AUC) for the subcutaneous (SC) injection to the AUC for the intravenous (IV) infusion, where AUC is assessed by plasma Rezafungin levels. Plasma rezafungin determined by LC-MS/MS methods.
Time Frame: Day 1 through Day 52
Population: The study was terminated on 27APR2020 due to safety concerns. No subjects were enrolled into any BA cohort.
Groups:
- BA 1: 100 mg (1 injection of 1.0 mL) or maximum tolerated dose (MTD) determined in SAD of Rezafungin administered subcutaneously into the abdomen on Day 1, and 100 mg (250 mL) or MTD of Rezafungin administered via intravenous infusion on Day 22 in an open label manner.
- BA 2: 100 mg (250 mL) or maximum tolerated dose (MTD) determined in SAD of Rezafungin administered via intravenous infusion on Day 1, and 100 mg (1 injection of 1.0 mL) or MTD of Rezafungin administered subcutaneously into the abdomen on Day 22 in an open label manner.
Arm/Group | BA 1 | BA 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days: from Day 1 (administration of first dose) to Day 30 (final study visit).
Description: AEs were defined according to ICH E6.
  Any medical condition present at the time of screening was considered baseline and was not reported as an AE. If the severity of any pre-existing medical condition increased, it was recorded as an AE.
Groups:
- SAD1: 1 mg (1 injection of 0.1 ml diluted 1:10 in 5% Dextrose Injection, USP) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=3 (no sentinel dosing) on Day 1 in a double-blind manner.
  Randomized 3:1.
- SAD2: 10 mg (1 injection of 0.1 ml) of Rezafungin administered subcutaneously into the abdomen as a single dose, n=6 (1 sentinel, 5 non-sentinel) on Day 1 in a double-blind manner.
  Randomized 3:1.
- SAD Placebo: Placebo participants across all SAD cohorts: 1 mg (1 injection of 0.1 ml diluted 1:10 in 5% Dextrose Injection, USP), 10 mg (1 injection of 0.1 ml), 30 mg (1 injection of 0.3 ml)
Arm/Group | SAD1 | SAD2 | SAD Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD1 (N=3) | SAD2 (N=6) | SAD Placebo (N=3)
Sinus bradycardia (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0) — SOC: General disorders and administration site conditions
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — SOC: General disorders and administration site conditions
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Basophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time shortened (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT04117607/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04117607/SAP_002.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT04117607/ICF_000.pdf